CLINICAL TRIAL: NCT01349517
Title: Health-related Quality of Life of Patients With Esophageal Cancer After Surgery in China: A Prospective Cohort Study From Multi-center
Brief Title: Health-related Quality of Life of Patients With Esophageal Cancer After Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: The First Hospital of Jilin University (Other); Fujian Medical University Union Hospital (Other); Shanxi Province Cancer Hospital (Other); Wuxi People's Hospital (Other); Linyi People's Hospital (Other)
Responsible Party: Tan Lijie MD, Associate Professor of Surgery, Zhong Shan Hospital, Fu Dan University, Shanghai, China,
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSchest2011001
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-01

CONDITIONS: Esophageal Cancer
Keywords: health-related quality of life(HRQL); Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MIE Group (Other): The patients in this group would perform minimal invasive three-incision subtotal esophagectomy (thoracoscopic and/or laparoscopic)
  Interventions: Procedure: MIE
- Three-incision esophagectomy group (Other): The patients in this group would perform three-incision subtotal esophagectomy (thoracotomy and laparotomy)
  Interventions: Procedure: Three-incision thoracotomy
- Ivor-Lewis esophagectomy group (Other): The patients in this group would underwent Ivor-Lewis esophagectomy
  Interventions: Procedure: Ivor-Lewis esophagectomy
- Sweet esophagectomy group (Other): The patients in this group would underwent Sweet esophagectomy.
  Interventions: Procedure: Sweet esophagectomy

INTERVENTIONS:
Procedure: MIE — The patients in this group would perform minimal invasive three-incision subtotal esophagectomy (thoracoscopic and/or laparoscopic)
  Other Names: esophagectomy
  Arms: MIE Group
Procedure: Three-incision thoracotomy — The patients in this group would perform three-incision subtotal esophagectomy (thoracotomy and laparotomy)
  Other Names: esophagectomy
  Arms: Three-incision esophagectomy group
Procedure: Ivor-Lewis esophagectomy — The patients in this group would underwent Ivor-Lewis esophagectomy
  Other Names: esophagectomy
  Arms: Ivor-Lewis esophagectomy group
Procedure: Sweet esophagectomy — The patients in this group would underwent Sweet esophagectomy.
  Other Names: esophagectomy
  Arms: Sweet esophagectomy group

SUMMARY:
The purpose of this multi-center prospective cohort study is to study the health-related quality of life (HRQL) together with other outcomes of patients with esophageal cancer after surgery in China.

DETAILED DESCRIPTION:
* To study the influence of health-related quality of life of patients with esophageal cancer before and after surgery.
* To compare the impact of different procedures on the the health-related quality of life of patients with esophageal cancer.
* To compare morbidities and oncological results(3,5- year survival) from different procedures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I/II esophageal cancer
* Normal blood test of basic metabolism panel
* Pulmonary function: FEV1 > 1.2L, FEV1% > 50%, DLCO > 50%
* Heart function: NY grade I and grade II

Exclusion Criteria:

* Mental disorders
* Combination with other cancers
* With a previous history of thoracic or ventral surgery

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | postoperative 2 year
  Health related quality of life from the different precedure groups (assessed by EORTC QLQ C-30 and OES-18)

SECONDARY OUTCOMES:
Morbidity Mortality Survival rate | 5 years
  * Perioperative morbidity and mortality from the different precedure groups.
  * 3-and 5-year survival rate between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Study Chair — Zhongshan Hospital, Fudan University, China
Locations (1):
- Zhong Shan Hospital, Fu Dan University, Shanghai, Shanghai Municipality, China